CLINICAL TRIAL: NCT00488514
Title: Study TXA107977, a Long-Term Safety Study of a Combination Product Containing Sumatriptan Succinate and Naproxen Sodium for the Treatment of Migraine in Adolescents
Brief Title: Long-Term Safety of Treximet (Sumatriptan/Naproxen Sodium) for Migraine in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXA107977
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2010-09-06 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2016-10

CONDITIONS: Migraine Disorders
Keywords: Long-term Safety; Migraine; Adolescent Migraine Headache; sumatriptan succinate; naproxen sodium
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Drug (Other): Combination Tablet of Treximet (sumatriptan/naproxen sodium)
  Interventions: Drug: Combination Tablet of Treximet (sumatriptan/naproxen sodium)

INTERVENTIONS:
Drug: Combination Tablet of Treximet (sumatriptan/naproxen sodium) — Combination Tablet of Treximet(sumatriptan/naproxen sodium)
  Other Names: Combination Product (sumatriptan succinate / naproxen sodium)

SUMMARY:
This study was designed to determine long-term safety of TREXIMET (sumatriptan/naproxen sodium) in adolescents for the acute treatment of migraine.

DETAILED DESCRIPTION:
This study was designed to determine long-term safety of TREXIMET (sumatriptan/naproxen sodium) in adolescents (aged 12 to 17 years) for the acute treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 12 and 17 years old at the Screening visit.
* If subject is female, she must have a negative urine pregnancy test at screening, does not plan to become pregnant during the course of the study and agrees to use an acceptable method of birth control (i.e., a method with a failure rate <1% or abstinence) if she is/becomes sexually active.
* Subject has migraine with or without aura (2004 ICHD-II criteria).
* Subject has history suggestive of typical migraine attacks with duration of about 2 or more hours (untreated, or unsuccessfully treated).
* Subject has at least 2, but not more than 8, migraine attacks per month in each of the 2 months prior to the Screening visit.
* Subject has at least a 6-month history of moderate to severe migraine attacks, sufficient to establish a definitive diagnosis of migraine.
* Subject is able to distinguish migraine from other headaches (e.g., tension-type headaches).
* Subject and subject's parent or legal guardian are willing and able to provide informed consent prior to entry into this treatment phase of the study.
* Subject and subject's parent or legal guardian are able to read and write English or Spanish.
* Subject is able to understand and complete the electronic device to report treatment information.

Exclusion Criteria:

* Subject is < 75 pounds (33.3kg).
* Subject has ≥15 headache days per month in total, retinal (ICHD-II 1.4), basilar (ICHD-II 1.26) or hemiplegic migraine (ICHD-II 1.25), or secondary headaches.
* Subject, in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease (See Appendix 1, section 11.1).
* Subject has uncontrolled hypertension (See Appendix 2, section 11.2) or is taking any angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker.
* Subject has a history of congenital heart disease, cardiac arrhythmias requiring medication, or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in this study.
* Subject has evidence or history of any ischemic vascular diseases including: ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome, or signs/symptoms consistent with any of the above.
* Subject has evidence or history of central nervous system pathology including stroke and/or transient ischemic attacks (TIAs), epilepsy or structural brain lesions which lower the convulsive threshold; or has been treated with an antiepileptic drug for seizure control within 5 years prior to screening.
* Subject has a history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study.
* Subject has hypersensitivity, allergy, intolerance, or contraindication to the use of any triptan, NSAID or aspirin (including all sumatriptan and naproxen preparations) or has nasal polyps and asthma.
* Subject is currently taking, or has taken in the previous three months, a migraine prophylactic medication containing methysergide or dihydroergotamine; or is taking a medication that is not stabilized (i.e., change of dose within the past 2 months) for either chronic or intermittent migraine prophylaxis or for a co-morbid condition that is not stabilized.
* Subject has a recent history of regular use of opioids or barbiturates for treatment of his/her migraine headache and/or other non-migraine pain. Regular use is defined as an average of 4 days per month over the last 6 months.
* Subject has taken, or plans to take, a monoamine oxidase inhibitor (MAOI), including herbal preparations containing St. John's Wort (Hypericum perforatum), anytime within the 2 weeks prior to screening through 2 weeks post final study treatment.
* Subject history of any bleeding disorder or is currently taking any anti-coagulant or any antiplatelet agent.
* Subject has evidence or history of any gastrointestinal surgery or GI ulceration or perforation in the past six months, gastrointestinal bleeding in the past year; or evidence or history of inflammatory bowel disease.
* Subject tests positive for illicit substances on toxicology screen, or has evidence of alcohol or substance abuse within the last year, or any concurrent medical or psychiatric condition which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this clinical trial.
* Subject has participated in an investigational drug trial within the previous 4 weeks or plans to participate in another study at any time during this study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 656 (Actual)
Dates: Start 2007-07-13; Primary Completion 2009-08-01 (Actual); Study Completion 2009-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (75):
- United States (75):
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Chico, California
  - GSK Investigational Site, Fair Oaks, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, East Hartford, Connecticut
  - GSK Investigational Site, Fairfield, Connecticut
  - GSK Investigational Site, Loxahatchee Groves, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Anderson, Indiana
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Murray, Kentucky
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Paw Paw, Michigan
  - GSK Investigational Site, Protage, Michigan
  - GSK Investigational Site, Richland, Michigan
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Ridgewood, New Jersey
  - GSK Investigational Site, Vorhees, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Amherst, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Mount Vernon, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Plainview, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Williamsville, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Westerville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Nassau Bay, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Bremerton, Washington
  - GSK Investigational Site, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] McDonald SA, Hershey AD, Pearlman E, Lewis D, Winner PK, Rothner D, Linder SL, Runken MC, Richard NE, Derosier FJ. Long-term evaluation of sumatriptan and naproxen sodium for the acute treatment of migraine in adolescents. Headache. 2011 Oct;51(9):1374-87. doi: 10.1111/j.1526-4610.2011.01965.x. Epub 2011 Jul 28. PMID 21797863
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: TXA107977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: TXA107977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TXA107977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TXA107977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TXA107977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TXA107977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TXA107977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- 85 mg Sumatriptan/500 mg Naproxen Sodium: Combination Tablet: 85 milligrams (mg) sumatriptan and 500 mg naproxen sodium. A single Combination Tablet was supplied for each migraine attack, not to exceed one tablet in 24 hours.
Period: Overall Study
Arm/Group | 85 mg Sumatriptan/500 mg Naproxen Sodium
Started | 656
Completed | 363
Not Completed | 293
Not completed — Adverse Event | 41
Not completed — Lost to Follow-up | 44
Not completed — Protocol Violation | 32
Not completed — Withdrawal by Subject | 106
Not completed — Lack of Efficacy | 28
Not completed — Did not meet criteria for treatment | 30
Not completed — Postive drug screen | 1
Not completed — Withdrawn per medical monitor decision | 2
Not completed — Investigator decision | 1
Not completed — Participant had too few migraines | 5
Not completed — Increase in number of migraines | 2
Not completed — Increased use of concomitant medication | 1

BASELINE CHARACTERISTICS:
Groups:
- 85 mg Sumatriptan/500 mg Naproxen Sodium: Combination Tablet: 85 milligrams (mg) sumatriptan and 500 mg naproxen sodium.
Arm/Group | 85 mg Sumatriptan/500 mg Naproxen Sodium
Number analyzed (Participants) | 622
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data were collected in the Safety Population, comprised of all participants in the Enrolled Population (all participants entered into the trial and categorized as "started" in the Participant Flow module) who took at least one dose of study drug.
  Years | 14.7 (1.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 367
  Male | 255
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 527
  Africian American | 71
  American Indian or Alaskan Native | 10
  Asian | 4
  African American/African Heritage and Asian | 2
  African American/African Heritage and White | 3
  American Indian or Alaskan Native and White | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Drug-related Adverse Events
Description: The number of participants with a drug-related adverse event (AE). Frequency threshold for reporting a drug-related AE: >=2% participants recorded as having at least one occurrence of a reported drug-related AE.
Time Frame: Baseline through End of Study (up to Month 12)
Population: Enrolled Population: all participants entered into the trial and dispensed the Combination Tablet, regardless of whether they ever took the Combination Tablet
Measure: Number; unit: participants
Groups:
- 6 Month Completer Population: Participants in the Enrolled Population who were treated with at least one dose of the combination tablet, completed at least one study visit (3- or 6-month visit), provided data for at least 6 migraines, and who continued in the study for at least 166 days
- 12 Month Completer Population: Participants in the Enrolled and 6 Month Completer Populations who completed at least one study visit in the second six-month period (9- or 12-month visit), provided data for at least 12 migraines, and who continued in the study for at least 346 days. The 12 Month Completer Population is a subset of those participants who completed or remained in the study for at least 346 days.
- Safety Population: Participants in the Enrolled Population who took at least one dose of the combination tablet
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | Safety Population
Number analyzed (Participants) | 333 | 181 | 622
participants
  At least one drug-related adverse event | 93 | 46 | 170
  Nausea | 19 | 11 | 44
  Dizziness | 7 | 3 | 20
  Muscle tightness | 10 | 5 | 18
  Chest discomfort | 10 | 3 | 16
  Paresthesia | 8 | 2 | 14
  Throat tightness | 11 | 6 | 14
  Somnolence | 9 | 2 | 14
  Neck pain | 6 | 3 | 12
  Flushing | 5 | 2 | 8

2. Secondary Outcome: Number of Participants With Any Adverse Event Categorized by Severity
Description: The number of participants with at least one mild (an event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities), moderate (an event that is sufficiently discomforting to interfere with normal everyday activities), or severe adverse event (an event that prevents normal everyday activities) was recorded.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | Safety Population
Number analyzed (Participants) | 333 | 181 | 622
participants
  Mild | 74 | 43 | 127
  Moderate | 140 | 72 | 220
  Severe | 24 | 14 | 44

3. Secondary Outcome: Number of Participants With Any Adverse Event Categorized Over Time
Description: The number of participants with an adverse event occurring in either the first six months of the study (months 0-6; <=194 days) or the second six months of the study (months 6-12; =>194 days until end of study) was recorded.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | Safety Population
Number analyzed (Participants) | 333 | 181 | 622
participants
  First six months of study | 208 | 112 | 348
  Second six months of study | 143 | 85 | 191

4. Secondary Outcome: Number of Participants With Any Adverse Event Categorized by Participant Age
Description: The number of participants with any adverse event by age group (12-14 and 15-17 years) is recorded.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | Safety Population
Number analyzed (Participants) | 333 | 181 | 622
participants
  Ages 12-14 | 104 | 57 | 175
  Ages 15-17 | 135 | 73 | 218

5. Secondary Outcome: Number of Participants With Any Adverse Event Categorized by Participant Race
Description: The number of participants with any adverse event was categorized by race. The category "Other" captures : American Indian or Alaskan Native; Asian, Native Hawaiian, or Other Pacific Islander; African American/African Heritage and Asian; African American/African Heritage and White; and American Indian or Alaskan Native and White.
Time Frame: Baseline through End of Study (up to Month 12)
Population: Safety Population: all participants in the Enrolled Population who took at least one dose of the combination tablet
Measure: Number; unit: participants
Arm/Group | 85 mg Sumatriptan/500 mg Naproxen Sodium
Number analyzed (Participants) | 622
participants
  Caucasian | 344
  African American | 35
  Other | 14

6. Secondary Outcome: Number of Participants With Any Adverse Event Categorized by Participant Gender
Description: The number of participants with adverse events by gender is recorded.
Time Frame: Baseline through End of Study (up to Month 12)
Population: Safety Population: all participants in the Enrolled Population who took at least one dose of the combination tablet
Measure: Number; unit: participants
Arm/Group | 85 mg Sumatriptan/500 mg Naproxen Sodium
Number analyzed (Participants) | 622
participants
  Female | 238
  Male | 155

7. Secondary Outcome: Number of Participants With Any Adverse Event That Occurred Within 3 or 5 Days of the First Dose of the Combination Tablet
Description: The number of participants with adverse events that occurred within 3 or 5 days of their first dose of the Combination Tablet was recorded.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | Safety Population
Number analyzed (Participants) | 333 | 181 | 622
participants
  Within 3 days | 66 | 35 | 128
  Within 5 days | 66 | 35 | 130

8. Secondary Outcome: Number of Tablets Taken, After Which at Least One Adverse Event Occurred Within 3 or 5 Days of Dosing With That Combination Tablet
Description: The number of events that occurred within 3 or 5 days of dosing with the combination tablet on a per tablet basis. A total of 8413, 5876, and 9989 tablets were taken by the 6 Month Completer, 12 Month Completer, and the Safety Populations, respectively.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 1
Measure: Number; unit: tablets
Groups:
- 6 Month Completer Population: Participants in the Enrolled Population who were treated with at least one dose of the combination tablet , completed at least one study visit (3- or 6-month visit), provided data for at least 6 migraines, and who continued in the study for at least 166 days
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | Safety Population
Number analyzed (Participants) | 333 | 181 | 622
tablets
  Number of tablets with an AE within 3 days | 917 | 667 | 1116
  Number of tablets with an AE within 5 days | 970 | 706 | 1178

9. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatinine, Potassium, and Blood Urea Nitrogen (BUN) Values of Interest That Shifted From Normal at Baseline to Abnormal at the End of Study Visit
Description: A shift from "normal to low," for example, indicates that a value was normal at baseline but low at the end of study visit. The value ranges were determined by the central laboratory. Reference ranges: ALT, 12 years old (y): 0-45 Units/liter (U/L), >13 y: 0-48 U/L; AST, 12 y: 0-42 U/L, >13 y 0-42 U/L; creatinine, 12 y: 27-88 micromoles/liter (UMOL/L), >13 y: 44-124 UMOL/L; potassium, 12 y: 3.5-5.5 millimoles/liter (MMOL/L), >13 y: 3.5-5.3 MMOL/L; BUN, 12-17 y: 24-101 milligrams (mg)/deciliter (dL).
Time Frame: Baseline through End of Study (up to Month 12)
Population: Enrolled Population: all participants entered into the trial and dispensed the Combination Tablet, regardless of whether they ever took the Combination Tablet. The number of participants with an assessment may vary, depending on the number of assessments completed at each visit.
Measure: Number; unit: participants
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | Safety Population
Number analyzed (Participants) | 330 | 179 | 565
participants
  ALT, normal to high, n=330, 179, 565 | 2 | 1 | 3
  ALT, normal to low, n=330, 179, 565 | 0 | 0 | 0
  AST, normal to high, n=329, 179, 562 | 1 | 1 | 3
  AST, normal to low, n=329, 179, 562 | 0 | 0 | 0
  Creatinine, normal to high, n=330, 179, 565 | 0 | 0 | 0
  Creatinine, normal to low, n=330, 179, 565 | 2 | 1 | 2
  Potassium, normal to high, n=329, 179, 562 | 1 | 0 | 4
  Potassium, normal to low, n=329, 179, 562 | 3 | 2 | 6
  BUN, normal to high, n=330, 179, 565 | 0 | 0 | 1
  BUN, normal to low, n=330, 179, 565 | 2 | 0 | 9

10. Secondary Outcome: Number of Participants With Hematocrit and Hemoglobin Values of Interest That Shifted From Normal at Baseline to Abnormal at the End of Study Visit
Description: A shift from "normal to low," for example, indicates that a value was normal at baseline but low at the end of study visit. The value ranges were determined by the central laboratory. Reference ranges: hemoglobin, 12-17 years old (y): 120-160 grams (g)/L; hematocrit (expressed as the percentage of blood occupied by red blood cells), 12-17 y: 0.360-0.490.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | Safety Population
Number analyzed (Participants) | 318 | 176 | 546
participants
  Hemoglobin, normal to high, n=318,176, 546 | 6 | 0 | 9
  Hemoglobin, normal to low, n=318,176, 546 | 10 | 6 | 20
  Hematocrit, normal to high, n=318,176, 546 | 2 | 0 | 4
  Hematocrit, normal to low, n=318,176, 546 | 17 | 10 | 29

11. Secondary Outcome: Mean Height for All Study Participants at the Indicated Time Points
Time Frame: Screening and Months 3, 6, 9, and 12
Population: Safety Population: all participants in the Enrolled Population who took at least one dose of the combination tablet. The number of participants with an assessment may vary by visit, depending on the number of assessments completed at each visit.
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- 12-14 Years: Participants who were 12-14 years old at the time of the Screening Visit
- 15-17 Years: Participants who were 15-17 years old at the time of the Screening Visit
- 12-17 Years: All participants in the Enrolled Population who took at least one dose of study drug
Arm/Group | 12-14 Years | 15-17 Years | 12-17 Years
Number analyzed (Participants) | 285 | 337 | 622
centimeters
  Screening, n=285, 337, 622 | 160.2 (9.15) | 167.0 (8.80) | 163.9 (9.57)
  Month 3, n=271, 308, 579 | 161.3 (9.09) | 167.3 (8.92) | 164.5 (9.48)
  Month 6, n=224, 249, 473 | 162.6 (9.12) | 167.3 (8.81) | 165.1 (9.26)
  Month 9, n=198, 221, 419 | 163.8 (8.92) | 167.6 (8.39) | 165.8 (8.84)
  Month 12, n=178, 198, 376 | 165.3 (8.86) | 167.9 (8.70) | 166.7 (8.86)

12. Secondary Outcome: Mean Weight for All Study Participants at the Indicated Time Points
Time Frame: Screening and Months 3, 6, 9, and 12
Population: Safety Population: all participants in the Enrolled Population who took at least one dose of the combination tablet. The number of participants with an assessment may vary, depending on the number of assessments completed at each visit.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | 12-14 Years | 15-17 Years | 12-17 Years
Number analyzed (Participants) | 285 | 337 | 622
kilograms
  Screening, n=285, 337, 622 | 57.02 (15.450) | 66.57 (16.824) | 62.19 (16.881)
  Month 3, n=270, 306, 576 | 58.01 (16.012) | 66.61 (16.921) | 62.58 (17.037)
  Month 6, n=223, 248, 471 | 60.20 (16.976) | 66.61 (16.864) | 63.57 (17.200)
  Month 9, n=197, 220, 417 | 61.24 (17.149) | 66.90 (17.169) | 64.23 (17.372)
  Month 12, n=178, 198, 376 | 62.92 (17.406) | 67.35 (17.952) | 65.25 (17.810)

13. Secondary Outcome: Mean Body Mass Index (BMI) for All Study Participants at the Indicated Time Points
Description: BMI = (Weight in kilograms)/(height in centimeters/100)^2
Time Frame: Screening and Months 3, 6, 9, and 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kilograms per meters squared
Arm/Group | 12-14 Years | 15-17 Years | 12-17 Years
Number analyzed (Participants) | 285 | 337 | 622
kilograms per meters squared
  Screening, n=285, 337, 622 | 22.01 (4.611) | 23.77 (5.249) | 22.97 (5.040)
  Month 3, n=270, 306, 576 | 22.09 (4.740) | 23.71 (5.267) | 22.95 (5.087)
  Month 6, n=223, 248, 471 | 22.54 (4.949) | 23.74 (5.455) | 23.17 (5.251)
  Month 9, n= 197, 220, 417 | 22.58 (4.904) | 23.74 (5.431) | 23.20 (5.215)
  Month 12, n=178, 198, 376 | 22.81 (4.969) | 23.79 (5.633) | 23.33 (5.345)

14. Secondary Outcome: Mean Blood Pressure for All Study Participants at the Indicated Time Points
Description: At each visit, a participant's blood pressure was taken three times. The average of the three readings was then calculated for each participant at each visit (mean blood pressure). The outcome measure represents the average of the mean blood pressure of all of the study participants. SBP, systolic blood pressure; DBP, diastolic blood pressure.
Time Frame: Screening and Months 3, 6, 9, and 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | 12-14 Years | 15-17 Years | 12-17 Years
Number analyzed (Participants) | 285 | 337 | 622
millimeters of mercury (mmHg)
  SBP, Screening, n=285, 337, 622 | 107.4 (10.08) | 110.2 (10.15) | 108.9 (10.21)
  SBP, Month 3, n=270, 308, 578 | 107.2 (10.67) | 111.1 (10.19) | 109.3 (10.58)
  SBP, Month 6, n=224, 249, 473 | 109.2 (10.37) | 112.0 (10.39) | 110.6 (10.46)
  SBP, Month 9, n=198, 221, 419 | 109.6 (10.55) | 112.7 (10.63) | 111.2 (10.69)
  SBP, Month 12, n=178, 198, 376 | 111.0 (10.78) | 112.1 (10.22) | 111.5 (10.49)
  DBP, Screening, n=285, 337, 622 | 66.2 (7.72) | 69.0 (7.24) | 67.7 (7.58)
  DBP, Month 3, n=270, 308, 578 | 65.7 (7.33) | 68.4 (7.84) | 67.1 (7.72)
  DBP, Month 6, n=224, 249, 473 | 66.1 (7.29) | 68.4 (7.68) | 67.3 (7.58)
  DBP, Month 9, n=198, 221, 419 | 65.6 (6.79) | 68.9 (7.30) | 67.3 (7.25)
  DBP, Month 12, n=178, 198, 376 | 66.6 (8.40) | 69.9 (7.35) | 68.3 (8.03)

15. Secondary Outcome: Mean Heart Rate for All Study Participants at the Indicated Time Points
Description: A sitting heart rate was measured once for each participant at each visit.
Time Frame: Screening and Months 3, 6, 9, and 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 12-14 Years | 15-17 Years | 12-17 Years
Number analyzed (Participants) | 284 | 336 | 620
beats per minute
  Screening, n=284, 336, 620 | 75.8 (11.58) | 73.0 (10.20) | 7.43 (10.93)
  Month 3, n=266, 305, 571 | 76.9 (11.57) | 75.6 (11.57) | 76.2 (11.58)
  Month 6, n=221, 247, 468 | 77.5 (10.87) | 75.4 (10.22) | 76.4 (10.57)
  Month 9, n=198, 221, 419 | 76.9 (11.43) | 75.4 (11.13) | 76.1 (11.28)
  Month 12, n=178, 198, 376 | 76.8 (12.17) | 74.7 (10.41) | 75.7 (11.31)

16. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram Findings at Screening and at the Final Visit as Assessed by the Investigator
Description: The number of participants with an electrocardiogram (ECG) status of normal, abnormal, clinically significant (CS), or not clinically significant (NCS), as determined by the Investigator, was reported. Specific definitions of ECG categorizations were not provided; investigators were expected to apply reasonable standards of clinical judgment. Normal, all ECG parameters within accepted normal ranges; abnormal, ECG finding(s) outside of normal ranges; CS, ECG with a CS abnormality that meets exclusion criteria; NCS, ECG with an abnormality not CS or meeting exclusion criteria per investigator.
Time Frame: Screening and Final Visit (up to Month 12)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | 12-14 Years | 15-17 Years | 12-17 Years
Number analyzed (Participants) | 284 | 337 | 621
participants
  Screening, normal, n=284, 337, 621 | 224 | 270 | 494
  Screening, abnormal, NCS, n=284, 337, 621 | 60 | 67 | 127
  Screening, abnormal, CS, n=284, 337, 621 | 0 | 0 | 0
  Final Visit, Normal, n=248, 294, 542 | 196 | 220 | 416
  Final Visit, abnormal, NCS, n=248, 294, 542 | 52 | 74 | 126
  Final Visit, abnormal, CS, n=248, 294, 542 | 0 | 0 | 0

17. Secondary Outcome: Number of Treated Migraine Attacks
Description: The number of migraine attacks eligible for evaluation, not associated with rescue medication use, or prohibited medications, was summarized. Rescue medication was additional medication taken within 24 hours of Combination Tablet. Prohibited medications: ergot, opioid, barbiturate, 5-HT1 agonist, long-acting non-steroidal anti-inflammatory drug (NSAID), short-acting NSAID-containing compound, analgesic, anti-emetic, monoamine oxidase inhibitors, St. John's Wort, angiotensin-converting enzyme inhibitor, Angiotensin II receptor blockers, anti-coagulant, anti-platelet.
Time Frame: Baseline through End of Study (up to Month 12)
Population: Intent-to-Treat (ITT) Population: all participants who took at least one dose of study drug and had at least one post-treatment migraine assessment
Measure: Number; unit: treated migraine attacks
Arm/Group | 85 mg Sumatriptan/500 mg Naproxen Sodium
Number analyzed (Participants) | 591
treated migraine attacks
  All Migraines | 8517
  Migraines Without Rescue Medication | 7791
  Migraines Without Rescue or Prohibited Medication | 7657

18. Secondary Outcome: Number of Treated Attacks Classified as Migraine Pain-Free (MPF) Within 24 Hours of Dosing With the Combination Tablet
Description: The number of migraine attacks eligible for evaluation, not associated with rescue medication use, and not associated with either rescue medication use or prohibited medications were counted. Migraine Pain Free was defined as the migraine attack ending <= 24 hours after the participant was dosed with the Combination Tablet.
Time Frame: Baseline through End of Study (up to Month 12)
Population: ITT Population: all participants who took at least one dose of study drug and had at least one post-treatment migraine assessment
Measure: Number; unit: treated migraine attacks
Arm/Group | 85 mg Sumatriptan/500 mg Naproxen Sodium
Number analyzed (Participants) | 591
treated migraine attacks
  All Migraines | 6400
  Migraines Without Rescue Medication | 6142
  Migraines Without Rescue or Prohibited Medication | 6052

19. Secondary Outcome: Number of Treated Attacks Classified as Migraine Pain-Free (MPF) Within 4 Hours of Dosing With a Combination Tablet
Description: The number of migraine attacks eligible for evaluation, not associated with rescue medication use, and not associated with either rescue medication use or prohibited medications were counted. Migraine Pain Free was defined as the migraine attack ending <= 4 hours after the participant was dosed with the Combination Tablet.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 18
Measure: Number; unit: treated migraine attacks
Arm/Group | 85 mg Sumatriptan/500 mg Naproxen Sodium
Number analyzed (Participants) | 591
treated migraine attacks
  All Migraines | 5076
  Migraines Without Rescue Medication | 5020
  Migraines Without Rescue or Prohibited Medication | 5017

20. Secondary Outcome: Number of Treated Attacks Classified as Migraine Pain-Free Within 4 Hours That Were Also Pain Free Within 2 Hours of Dosing With the Combination Tablet
Description: as for outcome 19
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 18
Measure: Number; unit: treated migraine attacks
Arm/Group | 85 mg Sumatriptan/500 mg Naproxen Sodium
Number analyzed (Participants) | 591
treated migraine attacks
  All Migraines | 3623
  Migraines Without Rescue Medication | 3598
  Migraines Without Rescue or Prohibited Medication | 3596

21. Secondary Outcome: Average Number of Headaches, Migraine Attacks, and Treated Migraine Attacks Per Month
Description: The average number of headaches (non-migraine and migraine attacks), migraine attacks, and treated migraine attacks per month was calculated for each participant, based on their time in the study. The outcome measure represents the average of the mean number of the headaches, migraine headaches, and treated migraines per month of the study participants in the 6 Month, 12 Month, and ITT Populations. A treated attack is defined as a migraine treated with the Combination Tablet.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events
Groups:
- ITT Population: Participants in the Enrolled Population who took at least one dose of the combination tablet and had at least one post-treatment migraine assessment
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | ITT Population
Number analyzed (Participants) | 333 | 181 | 591
events
  Headaches | 3.3 (2.19) | 3.9 (2.29) | 3.0 (2.49)
  Migraines | 2.2 (1.17) | 2.6 (1.09) | 1.8 (1.23)
  Treated migraine attacks | 1.9 (1.05) | 2.4 (0.97) | 1.5 (1.11)

22. Secondary Outcome: Number of Total Migraines Headaches and Migraines Treated With the Combination Tablet
Description: The total number of migraine headaches and the number of migraine headaches treated with the Combination Tablet during the study were summarized.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 1
Measure: Number; unit: migraine attacks
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | ITT Population
Number analyzed (Participants) | 333 | 181 | 591
migraine attacks
  Total Migraines | 8290 | 5851 | 9937
  Treated Migraines | 7318 | 5234 | 8517

23. Secondary Outcome: Number of Migraine Attacks Rated With the Indicated Pain Severity
Description: The number of migraine attacks treated at the mild, moderate, or severe intensity were counted. Pain severity was assessed by participants based on a scale of 0-3: 0=no pain, 1=mild, 2= moderate, 3=severe.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 1
Measure: Number; unit: treated migraine attacks
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | ITT Population
Number analyzed (Participants) | 333 | 181 | 591
treated migraine attacks
  No pain | 0 | 0 | 0
  Mild | 1373 | 1009 | 1619
  Moderate | 3555 | 2535 | 4132
  Severe | 2385 | 1686 | 2759

24. Secondary Outcome: Number of Treated Migraine Attacks With Photophobia, Phonophobia, Nausea, Neck Pain, Sinus Pain, and Vomiting
Description: The number of treated migraine attacks with the reported migraine-associated symptoms of photophobia, phonophobia, nausea, neck pain, sinus pain, and vomiting were counted. Photophobia: sensitivity to light; phonophobia: sensitivity to sound.
Time Frame: Baseline through End of Study (up to Month 12)
Population: as for outcome 1
Measure: Number; unit: treated migraine attacks
Arm/Group | 6 Month Completer Population | 12 Month Completer Population | ITT Population
Number analyzed (Participants) | 333 | 181 | 591
treated migraine attacks
  Photophobia | 5608 | 4064 | 6528
  Phonophobia | 5221 | 3725 | 6063
  Nausea | 3120 | 2173 | 3690
  Neck pain | 3050 | 2172 | 3540
  Sinus pain | 2052 | 1424 | 2428
  Vomiting | 555 | 375 | 682

25. Secondary Outcome: Mean Change From Baseline in the Migraine Specific Quality of Life (QOL) Questionnaire for Adolescents (MSQ-A) Score at Months 3, 6, 9, and 12
Description: The MSQ-A consists of 14 items measuring how migraines affect QOL: Role Function (RF)-Restrictive (items 1-7) and RF-Preventative (items 8-11), examining the degree to which performance of daily activities is limited or interrupted, respectively, by migraine; RF-Emotional (items 12-14, examining frustration/helplessness due to migraine). Dimensions (dim.) are scored independently. The 14 items are reverse coded onto a 1-6 scale; dim. are then created by summing specific item scores and transforming raw total score onto a 0-100 scale. For each dim., higher scores indicate better health status.
Time Frame: Baseline and Months 3, 6, 9, and 12
Population: Enrolled Population: all participants entered into the trial and dispensed the Combination Tablet, regardless of whether they ever took the Combination Tablet. Due to data collection and/or assignment of a collected assessment to a visit, the number of participants analyzed at a given visit could vary.
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | ITT Population | 12 Month Completer Population
Number analyzed (Participants) | 457 | 160
points on a scale
  Role restrictive, Month 3, n=457, 160 | 10.1 (1.145) | 9.0 (1.952)
  Role restrictive, Month 6, n=366, 160 | 10.5 (1.302) | 8.2 (1.972)
  Role restrictive, Month 9, n=315, 148 | 13.7 (1.475) | 9.0 (2.155)
  Role restrictive, Month 12, n=291, 153 | 15.7 (1.530) | 11.5 (2.117)
  Role preventative, Month 3, n=457, 160 | 7.9 (1.110) | 9.6 (1.974)
  Role preventative, Month 6, n=366, 160 | 6.8 (1.212) | 8.3 (1.890)
  Role preventative, Month 9, n=315, 148 | 9.4 (1.473) | 8.2 (2.234)
  Role preventative, Month 12, n=291, 153 | 9.8 (1.441) | 8.4 (1.959)
  Role emotional , Month 3, n=457, 160 | 7.1 (1.287) | 7.9 (2.223)
  Role emotional, Month 6, n=366, 160 | 6.6 (1.441) | 7.2 (2.136)
  Role emotional, Month 9, n=315, 148 | 10.5 (1.625) | 9.0 (2.411)
  Role emotional, Month 12, n=291, 153 | 11.4 (1.694) | 7.1 (2.461)

26. Secondary Outcome: Number of Participants Categorized by Response to Each of the 3 Global Satisfaction Questions From the Patient Perception Migraine Questionnaire-Revised (PPMQ-R) at the Screening Visit
Description: The PPMQ-R is a fully validated 32-item questionnaire assessing participant satisfaction with acute migraine medication and includes 3 questions that assess satisfaction with respect to efficacy, side effects, and overall satisfaction (i.e., How effective the medication is overall, side effects of the medication, overall satisfaction with the medication). Each item is rated on a 7-point scale ranging from "very satisfied" (1) to "very dissatisfied" (7).
Time Frame: Screening
Population: as for outcome 25
Measure: Number; unit: participants
Groups:
- ITT Population: Participants in the Enrolled Population who took at least one dose of the combination tablet drug and had at least one post-treatment migraine assessment
Arm/Group | ITT Population | 6 Month Completer Population | 12 Month Completer Population
Number analyzed (Participants) | 562 | 316 | 174
participants
  Overall Efficacy, Very Satisfied | 36 | 22 | 11
  Overall Efficacy, Satisfied | 163 | 102 | 54
  Overall Efficacy, Somewhat Satisfied | 192 | 113 | 72
  Overall Efficacy, Neutral | 67 | 30 | 15
  Overall Efficacy, Somewhat Dissatisfied | 49 | 23 | 12
  Overall Efficacy, Dissatisfied | 43 | 22 | 8
  Overall Efficacy, Very Dissatisfied | 12 | 4 | 2
  Side Effects, Very Satisfied | 135 | 89 | 50
  Side Effects, Satisfied | 166 | 87 | 50
  Side Effects, Somewhat Satisfied | 77 | 45 | 26
  Side Effects, Neutral | 127 | 69 | 36
  Side Effects, Somewhat Dissatisfied | 29 | 13 | 6
  Side Effects, Dissatisfied | 18 | 6 | 2
  Side Effects, Very Dissatisfied | 11 | 7 | 4
  Overall Treatment Satisfaction, Very Satisfied | 50 | 30 | 11
  Overall Treatment Satisfaction, Satisfied | 192 | 113 | 70
  Overall Treatment Satisfaction, Somewhat Satisfied | 164 | 94 | 56
  Overall Treatment Satisfaction, Neutral | 67 | 35 | 16
  Treatment Satisfaction, Somewhat Dissatisfied | 31 | 13 | 9
  Overall Treatment Satisfaction, Dissatisfied | 43 | 23 | 9
  Overall Treatment Satisfaction, Very Dissatisfied | 15 | 8 | 3

27. Secondary Outcome: Number of Participants Categorized by Response to Each of the 3 Global Satisfaction Questions From the Patient Perception Migraine Questionaire-Revised (PPMQ-R) at Month 12
Description: as for outcome 26
Time Frame: End of Study/Month 12
Population: as for outcome 25
Measure: Number; unit: participants
Groups:
- 6 Month Completer Population: Participant in the Enrolled Population who were treated with at least one dose of the combination tablet, completed at least one study visit (3- or 6-month visit), provided data for at least 6 migraines, and who continued in the study for at least 166 days
Arm/Group | ITT Population | 6 Month Completer Population | 12 Month Completer Population
Number analyzed (Participants) | 171 | 144 | 110
participants
  Overall Efficacy, Very Satisfied | 66 | 59 | 48
  Overall Efficacy, Satisfied | 75 | 63 | 46
  Overall Efficacy, Somewhat Satisfied | 20 | 16 | 12
  Overall Efficacy, Neutral | 7 | 5 | 3
  Overall Efficacy, Somewhat Dissatisfied | 2 | 1 | 1
  Overall Efficacy, Dissatisfied | 1 | 0 | 0
  Overall Efficacy, Very Dissatisfied | 0 | 0 | 0
  Side Effects, Very Satisfied | 55 | 49 | 42
  Side Effects, Satisfied | 61 | 51 | 40
  Side Effects, Somewhat Satisfied | 24 | 21 | 14
  Side Effects, Neutral | 11 | 10 | 6
  Side Effects, Somewhat Dissatisfied | 12 | 7 | 3
  Side Effects, Dissatisfied | 5 | 4 | 3
  Side Effects, Very Dissatisfied | 3 | 2 | 2
  Overall Treatment Satisfaction, Very Satisfied | 71 | 64 | 51
  Overall Treatment Satisfaction, Satisfied | 76 | 61 | 47
  Overall Treatment Satisfaction, Somewhat Satisfied | 13 | 10 | 6
  Overall Treatment Satisfaction, Neutral | 6 | 5 | 2
  Treatment Satisfaction, Somewhat Dissatisfied | 3 | 3 | 3
  Overall Treatment Satisfaction, Dissatisfied | 1 | 0 | 0
  Overall Treatment Satisfaction, Very Dissatisfied | 1 | 1 | 1

ADVERSE EVENTS:
Arm/Group | Safety Population | 6 Month Completer Population | 12 Month Completer Population
Serious Adverse Events (participants affected / at risk) | 4/622 | 3/333 | 1/181
Other Adverse Events (participants affected / at risk) | 257/622 | 159/333 | 89/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=622) | 6 Month Completer Population (N=333) | 12 Month Completer Population (N=181)
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1
Hemolytic anemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=622) | 6 Month Completer Population (N=333) | 12 Month Completer Population (N=181)
Nausea (Gastrointestinal disorders) | 55 | 28 | 16
Upper respiratory tract infection (Infections and infestations) | 54 | 39 | 22
Nasopharyngitis (Infections and infestations) | 48 | 35 | 20
Sinusitis (Infections and infestations) | 37 | 27 | 19
Dizziness (Nervous system disorders) | 25 | 10 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 24 | 12 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 16 | 10
Migraine (worsening) (Nervous system disorders) | 22 | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 16 | 10
Muscle tightness (Musculoskeletal and connective tissue disorders) | 20 | 12 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 13 | 7
Dysmenorrhoea (Reproductive system and breast disorders) | 19 | 14 | 12
Pyrexia (General disorders) | 14 | 12 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.